CLINICAL TRIAL: NCT06835387
Title: Phase II Study of NALIRIFOX (Nanoliposomal Irinotecan + Oxaliplatin With Fluorouracil and Folinic Acid) in Advanced Unresectable Small Bowel Tumors
Brief Title: Study of NALIRIFOX in Advanced Unresectable Small Bowel Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tiago Biachi de Castria (Other)
Collaborators: Ipsen (Industry); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor-Investigator, Tiago Biachi de Castria, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI23-617
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Small Bowel Adenocarcinoma
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: Subjects will receive treatment on Day 1 and Day 15 of each 28-day cycle consisting of the following: nanoliposomal irinotecan at 50 mg/m2, followed by oxaliplatin 60 mg/m2, followed by leucovorin at 400 mg/m2 30 minutes after completion of oxaliplatin, followed by 5-FU 2400 mg/m2 60 minutes after leucovorin completion. Patients will receive up to 6 cycles of NALIRIFOX then based on response and per physician discretion, de-escalated maintenance treatment with NALIRIFOX minus oxaliplatin may continue. Subjects will continue de-escalated maintenance treatment until progression per RECIST 1.1, intolerable toxicity or physician/subject choice to discontinue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NALIRIFOX and De-escalated maintenance (Experimental): Cycle 1 to Cycle 6: NALIRIFOX Subjects will receive treatment on Day 1 and Day 15 of each 28-day cycle consisting of the following: nanoliposomal irinotecan at 50 mg/m2, followed by oxaliplatin 60 mg/m2, followed by leucovorin at 400 mg/m2 30 minutes after completion of oxaliplatin, followed by 5-FU 2400 mg/m2 60 minutes after leucovorin completion. Patients will receive up to 6 cycles of NALIRIFOX.
  Cycle 7+: De-escalated Maintenance:
  Based on response to Cycles 1-6 and per physician discretion, de-escalated maintenance treatment with NALIRIFOX minus oxaliplatin may continue as de-escalated maintenance treatment until progression per RECIST 1.1, intolerable toxicity or physician/subject choice to discontinue.
  Interventions: Drug: Nanoliposomal irinotecan; Drug: Oxaliplatin; Drug: 5 fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Nanoliposomal irinotecan — Nanoliposomal Irinotecan 50 mg/m2 will be administered over 90 minutes (± 10 minutes) IV. All subjects must be pre-medicated prior to nanoliposomal irinotecan infusion with standard doses of dexamethasone and a 5-HT3 antagonist, or equivalent other anti-emetics (according to standard institutional practices).
  Other Names: Onivyde
Drug: Oxaliplatin — Oxaliplatin 60 mg/m2 will be administered over 120 minutes (± 10 minutes) IV. Institutional standards may be used for all aspects of oxaliplatin administration including premedication administration.
  Other Names: Eloxatin
Drug: 5 fluorouracil — 5-FU will be administered as a continuous infusion over 46 hours. Subjects will go home with an infusion pump and return to clinic at the end of infusion for removal of the pump or, if possible, the pump may be removed at the subject's home (except on Cycle 1 Day 3).
  Other Names: Tolak; Efudex; Fluoroplex
Drug: Leucovorin — Leucovorin 400 mg/m2 will be administered over 30 minutes IV.
  Other Names: Wellcovorin; folinic acid

SUMMARY:
The study regimen will be administered on an outpatient basis and all medications are administered intravenously (IV). Subjects will receive treatment on Day 1 and Day 15 of each 28-day cycle consisting of the following: nanoliposomal irinotecan at 50 mg/m2, followed by oxaliplatin 60 mg/m2, followed by leucovorin at 400 mg/m2 30 minutes after completion of oxaliplatin, followed by 5-FU 2400 mg/m2 60 minutes after leucovorin completion. Subjects will receive up to 6 cycles of NALIRIFOX then based on response and per physician discretion, de-escalated maintenance treatment with NALIRIFOX minus oxaliplatin may continue. Subjects will continue de-escalated maintenance treatment until progression per RECIST 1.1, intolerable toxicity or physician/subject choice to discontinue.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has been informed about the nature of the study, and has agreed to participate in the study, and signed the ICF prior to participation in any study-related activities. Also, as determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of ≤ 1 within 28 days prior to registration and within 7 days prior to start of study regimen.
4. Histological or cytologically confirmed small bowel adenocarcinoma per AJCC, 9th edition that has not been previously treated in the metastatic setting. Subjects treated in the adjuvant setting who completed treated > 6 months and do not have residual toxicities > Grade 1 are eligible. NOTE: Subjects with only localized disease or disease which will likely become resectable after chemotherapy (per investigator discretion) are NOT eligible.
5. Mismatch repair proficient (MMRp) and/or microsatellite stable (MSS) disease per institutional standard of care testing.
6. Subject has one or more metastatic lesions measurable by CT scan (or MRI, if the subject

   a. is allergic to CT contrast media) according to RECIST Version 1.1 criteria. Lesions in a prior radiation field must have progressed subsequent to radiotherapy to be considered measurable.
7. Demonstrate adequate organ function as defined below. All screening labs to be obtained within 28 days prior to registration and repeated within 7 days prior of C1D1.

   * Platelets (Plt) ≥ 100,000 cells/mm3
   * Absolute Neutrophil Count (ANC) ≥ 1,500 cells/mm3; without the use of hemopoietic growth factors
   * Hemoglobin (Hgb) ≥ 9 g/dL
   * Calculated creatinine clearance ≥ 30 mL/min; Cockcroft-Gault formula for actual body weight should be used for calculation. For subjects with a body mass index (BMI) > 30 kg/m2, adjusted body weight should be used instead
   * Total bilirubin ≤ 1.5 × ULN
   * Aspartate aminotransferase (AST) ≤ 2 × ULN; < 5× with liver metastases
   * Alanine aminotransferase (ALT) ≤ 2 × ULN; < 5× with liver metastases
   * Albumin ≥ 2.5 gm/dL
   * PT and PTT ≤ 1.5 x ULN; subjects on warfarin or other vitamin K antagonists should be discussed with the sponsor-investigator.
   * Urinalysis: Urinalysis results without clinically significant abnormalities, per the investigator's assessment
8. Electrocardiogram (ECG) without any clinically significant findings (QT interval corrected by Fridericia's formula (QTcF) ≤450 msec and no known arrhythmias) and per the investigator's assessment.
9. Females of childbearing potential must have a negative urine or serum pregnancy test within ≤ 7 days prior to registration. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from penile-vaginal intercourse or use an effective method(s) of contraception. Males able to father a child who are sexually active with a female of childbearing potential must be willing to abstain from penile-vaginal intercourse or use an effective method(s) of contraception.
11. Subjects infected with human immunodeficiency virus (HIV) are eligible if they meet all the following criteria:

    * CD4 count is ≥350 cells/uL, viral load is undetectable, and not taking prohibited cytochrome (CYP)-interacting medications;
    * Probable long-term survival with HIV if cancer were not present;
    * Stable on a highly active antiretroviral therapy (HAART) regimen for ≥ 4 weeks and willing to adhere to their HAART regimen with minimal overlapping toxicity and drug-drug interactions with the experimental agents in this study;
    * HIV is not multi-drug resistant;
    * Taking medication and/or receiving antiretroviral therapy that does not interact or have overlapping toxicities with the study medication.

    NOTE: Testing is not required at screening unless mandated by local policy.
12. Subjects with known chronic hepatitis B virus (HBV) infection, must have an undetectable HBV viral load on suppressive therapy, if indicated. Subjects with a history of hepatitis C virus (HCV) infection must have been treated and cured. For subjects with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial. NOTE: Testing is not required at screening unless mandated by local policy.

Exclusion Criteria:

1. Adenocarcinoma originating in the ampulla or appendix (duodenal tumors that involve the ampulla but originate in the duodenum are eligible).
2. Neuroendocrine or any other histology different than adenocarcinoma.
3. Prior treatment with irinotecan.
4. Prior treatment of SBA in the metastatic setting with surgery, radiotherapy, chemotherapy or investigational therapy:

   * Palliative radiotherapy is permitted but lesions in a prior radiation field must have progressed subsequent to radiotherapy to be considered measurable.
   * Placement of biliary stent/tube is permitted.
5. Known history of central nervous system (CNS) metastases. (subjects on a stable or decreasing dose of steroids and deemed clinically stable as per the investigator's assessment are eligible).
6. Clinically significant gastrointestinal disorder including hepatic disorders, bleeding, inflammation, occlusion, diarrhea > Grade 1, malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, or partial bowel obstruction.
7. Pregnant or breastfeeding. NOTE: breast milk cannot be stored for future use while the mother is being treated on study.
8. History of any second malignancy in the last 2 years; subjects with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible. Subjects with a history of other malignancies are eligible if they have been continuously disease free for at least 2 years prior to screening. Subjects who have a concurrent malignancy that is clinically stable and does not require tumor-directed treatment are eligible.
9. Known hypersensitivity to any of the components of nanoliposomal irinotecan, other liposomal products, or any components of 5-FU, LV or oxaliplatin.
10. Concurrent illnesses that would be a relative contraindication to trial participation such as active cardiac or liver disease, including:

    * Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before screening
    * High cardiovascular risk, including, but not limited to, recent coronary stenting or myocardial infarction in the past year prior to screening
    * New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure
11. Active infection or an unexplained fever >38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, subjects with tumor fever may be enrolled), which in the investigator's opinion might compromise the subject's participation in the study or affect the study outcome.
12. Major surgery, other than diagnostic surgery, within 4 weeks prior to consent.
13. Use of strong inhibitors or inducers of CYP3A, CYP2C8 and UGT1A1. Subjects are ineligible if:

    * they are unable to discontinue the use of strong inhibitors of CYP3A, CYP2C8 and UGT1A1 at least 1 week prior to consent;
    * they are unable to discontinue the use of strong CYP3A and CYP2C8 inducers at least 2 weeks prior to consent;
14. There is presence of any contraindications outlined in the Contraindications or Warnings and Precautions sections of the IB for nanoliposomal irinotecan, or in the prescribing information for 5-FU, LV or oxaliplatin.
15. Subjects who, in the opinion of the investigator, have symptoms or signs suggestive of clinically unacceptable deterioration of the primary disease at the time of screening.
16. History of systemic connective tissue disorders (e.g. lupus, scleroderma, arteritis nodosa).
17. Subjects who have received a live vaccine within 4 weeks prior to consent.
18. History of the following: interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies, and peripheral artery disease (e.g. claudication, Leo Buerger's disease).
19. Known low or absent dihydropyridine dehydrogenase (DPD) activity. This is not mandatory but where required by local regulations, testing for DPD deficiency must be performed using a validated method which is recommended by local health authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  ORR is defined as the proportion of subjects with a confirmed complete or partial response to treatment according to RECIST 1.1, by local assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  OS is defined as the time from initiation of study regimen to date of death due to any cause.
Time to Progression (TTP) | 3 years
  TTP is defined as the time from initiation of study regimen to date of disease progression by RECIST 1.1.
Duration of Response (DOR) | 3 years
  DOR is defined as the time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD (per RECIST 1.1) or ro death due to any cause, whichever comes first.
Number of Participants with Adverse Events | 3 years
  Adverse events will be assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Biachi de Castria, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Virginia Commonwealth University, Richmond, Virginia